CLINICAL TRIAL: NCT00552643
Title: Study to Evaluate Polyheal-1 in Treatment of Recalcitrant Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Polyheal Ltd. (Industry)
Responsible Party: Jordan Rubinson, CEO, Polyheal Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PH1-07-01
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Wounds and Injuries
Keywords: Recalcitrant ulcers; Chronic wounds; Venous insufficiency wounds; Ulcers; Exposed bones; Exposed Tendons; Granulation tissue; Polyheal 1; Wound care; Wound healing; Diabetic wounds healing; Post trauma; Post surgery complication; Recalcitrant wounds including venous, post-operative and post-traumatic chronic wounds with different etiologies including wounds with exposed bone and tendon.
MeSH Terms: conditions — Wounds and Injuries; Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Treatment with Polyheal 1
  Interventions: Device: Suspension of polystyrene beads (POLYHEAL 1)
- 2 (Active Comparator): Saline
  Interventions: Device: Saline (0.9% NaCl)

INTERVENTIONS:
Device: Suspension of polystyrene beads (POLYHEAL 1) — Topical application of Polyheal 1 (15 mL/200cm2 of wound area, TID, 28 days, one cycle
  Arms: 1
Device: Saline (0.9% NaCl) — Saline topical application 15 mL/200cm2 of wound area, TID, 28 days, one cycle
  Other Names: Physiological solution; 0.9% NaCl
  Arms: 2

SUMMARY:
The objective of this study is to evaluate the performance of Polyheal-1 compared to Saline in the treatment of recalcitrant wounds including venous, post-operative and post-traumatic chronic wounds with different etiologies including wounds with exposed bone and/or tendons.

DETAILED DESCRIPTION:
Chronic ulcers affect millions of people, and are a growing clinical problem seen most frequently in the elderly. Non-healing or slow healing wounds represent a major health burden and drain on resources, contributing to substantial disability, morbidity, and cost. Wound healing involves a well-orchestrated, complex process leading to repair of injured tissues. Basic principles of good wound care involve removal of necrotic tissue by mechanical, surgical or enzymatic debridement, wound bed preparation, and treatment of infection. In general, wounds that are being appropriately managed show measurable progress within 2-4 weeks. However despite delivering good wound care that includes providing the right dressings, nutritional support, topical care, and offering top-of-the-line support surfaces, wounds often become stagnated. Wounds refractory to treatment for 2-4 weeks are dubbed recalcitrant. Such wounds need sometime some stimuli to start the healing cascade. Polyheal-1, is thought do be potentially useful in triggering the healing process and can be particularly beneficial in stimulating the granulation process in chronic wounds of different etiologies e.g. venous, diabetic wounds, decubitus ulcers and post trauma/surgery complicated wounds. For instance exposed bones and tendons that are particularly difficult to be treated, were previously demonstrated to benefit from stimulation of granulation coverage by application of Polyheal 1.

In this protocol we intent to perform comparative study aimed at comparing performance of Polyheal I to Saline in treatment of recalcitrant wounds of different etiology such as venous and various post-operative wounds including cases were the exposed bone needs granulation coverage. Furthermore, patients with post- operative surgical complications such as sternum or partial foot amputation in diabetic patients will also be a subject of present investigation. Polyheal 1 will be compared to saline as this is the most commonly used treatment intended at keeping the wound moist and enabling progress of granulation and epithelization.

ELIGIBILITY:
Inclusion Criteria:

* The patient is 18 years of age and older.
* The patient has at least one recalcitrant wound (venous insufficiency, post- operative and post-traumatic chronic wounds with different etiology including those with open wounds) refractive to healing at least 4 weeks prior to treatment
* Patients defined as grade 4 or below on the granulometer including wounds with exposed bone or tendon.
* Patients will be eligible to participate in the study if their target lesion area of the edges is larger than 15cm2 and smaller than 200 cm2 at baseline in the group A of wounds caused by venous insufficiency or larger than 2cm2 and smaller than 200 cm2 at baseline in the group B of post-operative and post- traumatic chronic wounds with exposed bone, tendon and/or ligaments.
* The patient is expected to be available for the 12 weeks study.

Exclusion Criteria:

* Clinically significant arterial vascular disease with ABI index <0.45 if the peripheral pulse is not palpable.
* Wound has necrotic tissue which covers more than 50% of the wound area.
* Neuropathic wounds of diabetic origin.
* Roentgenic (X-ray) evidence of osteomyelitis in target wound in case that the bone is detectable by insertion of wire.
* Diabetic patients with HbA1c >11%
* Presence of a systemic infection or significant local infection such as cellulites, purulent drainage, gangrene, or necrosis at the target wound site, as well as nonviable tissue, sinus tracts or tunnels that cannot be removed by debridement.
* Previous history of any illness or condition that may impair wound healing, immune deficiency or connective tissue disease (e.g., SLE, AIDS), neurological disease (e.g., multiple sclerosis), dialysis due to renal disease and active hepatic disease.
* Patient is receiving, or has received within one month prior to Visit 1 any treatment known to impair wound healing, including but not limited to: corticosteroids, immuno- suppressive drugs, cytotoxic agents, radiation therapy and chemotherapy.
* Patient has a history of alcohol or drug abuse within the last two years.
* Presence or suspicion of any malignancy.
* Treatment with a dressing containing growth factors or other biological dressings within 15 days, prior to the screening visit.
* Female patients who are pregnant or nursing, or of childbearing potential and are not using adequate contraception.
* Participation in another clinical trial within 30 days prior to the Screening Visit or during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measures:The primary endpoint will be achievement of at least 75% light red granulation tissue, (grade 7 or 8 on the granulometer), | 12 weeks

SECONDARY OUTCOMES:
(1) time to complete wound closure measured in weeks, (2) achievement of complete wound closure, measured by number of patients out of total. (3) time to full bone coverage by granulation tissue measured in weeks. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gavriel Zeilig, DM, Principal Investigator — Sheba Medical Center
Locations (6):
- Israel (6):
  - Soroka University Medical Center, Beersheba
  - Hadassah Ein-Kerem Hospital, Jerusalem
  - Western Galilee Hospital, Nahariya
  - Sourasky Medical Center, Tel Aviv
  - High Risk Foot Clinic - Maccabi Health Services, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky